CLINICAL TRIAL: NCT04082442
Title: Evolocumab in Patients With Acute Myocardial Infarction: A Double-blind, Prospective, Randomized Placebo-Controlled Study
Brief Title: Evolocumab in Patients With Acute MI
Acronym: EVACS II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00206305
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Experimental): 420 mg evolocumab administered subcutaneously using an autoinjector/pen in ACS patients.
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously using an autoinjector/pen in ACS patients .
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Evolocumab — 420 mg evolocumab.
  Arms: Evolocumab
Drug: Placebos — Matching placebo.
  Arms: Placebo

SUMMARY:
Vascular and myocardial inflammation are significantly increased in Acute Coronary Syndrome (ACS) patients, are closely correlated to LDL-C levels, and are associated with these adverse consequences in the post-ACS patient population. Serum proprotein convertase subtilisin/kerin type 9 (PCSK9) levels are also increased in ACS, may raise LDL-C, and the investigators' pre-clinical studies indicate that PCSK9 is also a potent inducer of vascular inflammation. The addition of the PCSK9 antibody evolocumab, currently approved to lower LDL-C in certain patient populations, to current medical therapies would appear to be of particular benefit in patients with an ACS by markedly reducing LDL-C, stabilizing vulnerable plaque, and limiting inflammation-associated myocardial cell loss and resultant dysfunction.

DETAILED DESCRIPTION:
Despite aggressive early intervention and current secondary prevention strategies, many patients who survive hospitalization for an acute coronary syndrome (ACS) experience subsequent unfavorable outcomes, including recurrent ischemic events and unfavorable cardiac remodeling associated with progressive left ventricular dysfunction and congestive heart failure. Vascular and myocardial inflammation are significantly increased in ACS patients, are closely correlated with LDL-C levels, and are associated with these adverse consequences. Serum proprotein convertase subtilisin/kerin type 9 (PCSK9) levels are also increased in patients with ACS, may raise LDL-C, and the investigators' pre-clinical studies indicate that PCSK9 is also a potent inducer of vascular inflammation. The addition of evolocumab to current medical therapies may therefore be of particular benefit in these patients, by markedly reducing LDL-C, stabilizing vulnerable plaque, and limiting inflammation-associated myocardial cell loss and resultant dysfunction.

In this study, the investigators propose to test the effects of PCSK9 inhibition with evolocumab on LDL-C reduction, vascular and myocardial inflammation, cardiac function, and clinical outcomes in an ACS patient cohort.

The investigators propose a double-blind randomized study of 100 patients presenting with an ACS (ST-Elevation- and Non-ST-elevation myocardial infarction). One hundred ACS patients will be randomized to evolocumab, 420 mg or to placebo (50 in each group) during early hospitalization and will also receive current guideline-directed ACS therapy. Lipid profiles, including LDL-cholesterol levels, and traditional and novel serum markers of inflammation and endothelial function will be measured at presentation, during the index hospitalization, and at 30-day and six-month follow-up. Positron Emission Tomography (PET) scans to measure myocardial and vascular inflammation and echocardiograms will be performed during the early post-infarction period and at thirty days (PET and echocardiogram) and six-month (echocardiogram) following randomization. Clinical outcomes, such as angina class, will also be collected at the six-month follow-up visit.

The protocol and the primary and secondary lipid and inflammatory outcomes in this study are identical to those in NCT03515304 and therefore the data in the two studies may be analyzed together.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 90 years.
2. ST elevation myocardial infarction, with compatible symptoms and ECG changes.
3. Non ST elevation myocardial infarction, with a troponin I > 5ng/mL and with compatible symptoms and ECG changes.
4. Permission of attending physician.
5. Ability to understand the risk, benefits, and alternatives of participation.

Exclusion Criteria:

1. Scheduled for cardiac surgery.
2. Current treatment with a PCSK9 antibody.
3. Current participation in an intervention clinical trial.
4. Latex allergy
5. Previous adverse reaction to monoclonal antibodies
6. Non-English speaking
7. Female of childbearing potential. This is a female subject who has not used acceptable method(s) of birth control (see below) for at least one month prior to screening, unless the subject is sterilized or postmenopausal. Menopause is defined as: 12 months of spontaneous and continuous amenorrhea in a female > 55 year of age.

   * Acceptable method(s) of birth control definition: One highly effective method (methods that can achieve a failure rate of less than 1% per year when used consistently and correctly)

     * Combined hormonal (estrogen and progestogen) contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
     * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
     * Intrauterine device (IUD)
     * Intrauterine hormone-releasing system (IUS)
     * Bilateral tubal occlusion
     * Vasectomized partner
     * Sexual abstinence
8. Subject likely not to be available to complete all protocol-related study visits or procedures.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Leucker, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziogos E, Vavuranakis MA, Harb T, Foran PL, Blaha MJ, Jones SR, Lai S, Gerstenblith G, Leucker TM. Lipoprotein(a) concentrations in acute myocardial infarction patients are not indicative of levels at six month follow-up. Eur Heart J Open. 2023 Apr 5;3(2):oead035. doi: 10.1093/ehjopen/oead035. eCollection 2023 Mar. PMID 37095769
- [Derived] Vavuranakis MA, Jones SR, Ziogos E, Blaha MJ, Williams MS, Foran P, Schindler TH, Lai S, Schulman SP, Gerstenblith G, Leucker TM. The Trajectory of Lipoprotein(a) During the Peri- and Early Postinfarction Period and the Impact of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibition. Am J Cardiol. 2022 May 15;171:1-6. doi: 10.1016/j.amjcard.2022.01.058. Epub 2022 Mar 21. PMID 35314069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evolocumab | Placebo
Started | 50 | 50
Completed | 27 | 29
Not Completed | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evolocumab | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 61 (11) | 61.94 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 36 | 34 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 48 | 50 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 14 | 32
  White | 29 | 29 | 58
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL-Cholesterol
Description: The difference, in the percent change in LDL-cholesterol (mg/dL), from baseline to the 25-30 day values.
Time Frame: Baseline, 25-30 days
Measure: Mean (95% Confidence Interval); unit: percent change mg/dL
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 27 | 29
percent change mg/dL | -70.59 [-82 to -58.21] | -44.78 [-58.43 to -6.34]
Statistical Analysis 1: Comparison: Evolocumab vs Placebo; Test type: Superiority; p = .0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: FDG-PET Imaging Analysis of Inflammation as Mean Standardized Uptake Value (SUV)
Description: The change between early infarction period and thirty day assessments of PET-FDG assessed myocardial inflammation. A higher SUV value= worse inflammation. There are no standard values for this, since this study is the first to describe this in this patient population.
Time Frame: Baseline, 30 days
Population: participants who completed the follow-up scan at 30 days
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value (SUV)
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 11 | 14
Standardized Uptake Value (SUV) | -26.21 (22.61) | -14.52 (36.92)
Statistical Analysis 1: Comparison: Evolocumab vs Placebo; Test type: Superiority; p = .34, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days
Arm/Group | Evolocumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 5/50
Other Adverse Events (participants affected / at risk) | 4/50 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=50) | Placebo (N=50)
Angina (Cardiac disorders) | 2 | 2
Heart Failure (Cardiac disorders) | 0 | 1
PEA Arrest (Cardiac disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=50) | Placebo (N=50)
Episode of NSVT (Cardiac disorders) | 1 | 0
Atrial fibrilation (Cardiac disorders) | 0 | 1
Recurrent Ischemia (Cardiac disorders) | 1 | 0
Dyspepsia and constipation (Gastrointestinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Food related allergy (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04082442/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04082442/SAP_001.pdf